CLINICAL TRIAL: NCT02988453
Title: Mentalization-based Training for Adolescents With Conduct Disorder (MBT-CD): A Feasibility and Pilot Study
Brief Title: Mentalization-based Training for Adolescents With Conduct Disorder (MBT-CD)
Acronym: MBT-CD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: Heidelberg University, Psychotherapy Research Department (Unknown); Heidelberg University, Clinic for Child and Youth Psychiatry (Unknown); Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Svenja Taubner, Prof. Dr., Heidelberg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23011229
Record Dates: First submitted 2016-11-30; First posted 2016-12-09 (Estimated); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Conduct Disorder
Keywords: mentalization-based treatment; conduct disorder; adolescents
MeSH Terms: conditions — Conduct Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MBT-CD (Experimental): Mentalization-based treatment program
  Interventions: Other: MBT-CD

INTERVENTIONS:
Other: MBT-CD — MBT-CD is a disorder-specific modification of MBT, initially developed for patients with Borderline Personality Disorder. It is a manualized and psychodynamically oriented psychotherapy with the aim to increase the mentalization capacity of adolescents in close relationships. The therapy consists of 2 psychoeducational group sessions, 30 individual therapy sessions and 10 family sessions. The average duration of therapy is 6 months.

SUMMARY:
A feasibility and pilot trial to investigate the feasibility of a newly manualized psychotherapy "Mentalization-Based Training for Adolescents with Conduct Disorder (MBT-CD)"

DETAILED DESCRIPTION:
Background: Conduct Disorder is a severe and complex mental disorder with the highest incidence in adolescence. Previous studies have shown that family-oriented interventions are effective in the treatment of Conduct Disorder. However, most therapies focus rather on symptom management and less on etiological causes without inclusion of the family in the therapeutic process. Previous research has linked specific symptoms of Conduct Disorder with deficits in mentalization ability. Mentalization is the ability to perceive one's own and other's behavior as the product of affective and cognitive mental states. Low or missing mentalization abilities are regarded as a risk factor for the development and chronification of Conduct Disorder.

Aims: The study aims to investigate the feasibility of a newly manualized psychotherapy "Mentalization-Based Training for Adolescents with Conduct Disorder (MBT-CD)" that strives to decrease symptoms associated with Conduct Disorder by increasing mentalization in adolescents and their families.

Methods: The study is feasibility and piolot trial, carried out in Heidelberg (Germany), and Mainz (Germany). Adolescents aged between 11-18, who meet the DSM-5 criteria for Conduct Disorder will receive MBT-CD. Times of measurement: t0 (Screening), T1 (Baseline, at the beginning of therapy), T2 (3 months after the beginning of therapy), T3 (at the end of therapy, after 6 months), T4 (follow-up, after 9 months).

ELIGIBILITY:
Inclusion Criteria:

* main diagnosis conduct disorder (DSM-5 312.81,312.82)
* written informed consent

Exclusion Criteria:

* acute substance dependence
* sexual offenses
* acute psychotic symptoms, early or early-onset schizophrenia
* neurological impairments and low intelligence (IQ <80)
* non-German-speaking
* other clinical contra indication for outpatient psychotherapy (e.g. acute suicidality)

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2016-12; Primary Completion 2021-10 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Structured Clinical Interview for DSM-IV Axis II Disorders (SCID-II) | Change from baseline in SCID-II at 12 months (at the end of therapy)
Subtypes of Antisocial Behaviour Questionnaire (STAB) | Change from baseline in STAB at 6 months
Subtypes of Antisocial Behaviour Questionnaire (STAB) | Change from baseline in STAB at 12 months (at the end of therapy)
Subtypes of Antisocial Behaviour Questionnaire (STAB) | Change from baseline in STAB at 18 months (follow-up)
Reactive-Proactive-Aggression Questionnaire (RPQ) | Change from baseline in RPQ at 6 months
Reactive-Proactive-Aggression Questionnaire (RPQ) | Change from baseline in RPQ at 12 months (at the end of therapy)
Reactive-Proactive-Aggression Questionnaire (RPQ) | Change from baseline in RPQ at 18 months (follow-up)

SECONDARY OUTCOMES:
Global Assessment of Functioning (GAF) | Change from baseline in GAF at 12 months (at the end of therapy)
Clinical Global Impression (CGI-SI) | Change from baseline in CGI-SI at 12 months (at the end of therapy)
Levels of Personality Functioning - Questionnaire Adolescence (LoPF-QA) | Change from baseline in LoPF-QA at 12 months (at the end of therapy)
Levels of Personality Functioning - Questionnaire Adolescence (LoPF-QA) | Change from baseline in LoPF-QA at 18 months (follow-up)
Reflective Functioning Questionnaire (RFQ) | Change from baseline in RFQ at 12 months (at the end of therapy)
Reflective Functioning Questionnaire (RFQ) | Change from baseline in RFQ at 18 months (follow-up)
Movie for the Assessment of Social Cognition (MASC) | Change from baseline in MASC at 12 months (at the end of therapy)
10 round Trust Game Task (TGT) | Change from baseline in TGT at 12 months (at the end of therapy)
Social Hierarchy Task (SHT) | Change from baseline in SHT at 12 months (at the end of therapy)
Approach-Avoidance Task (AAT) | Change from baseline in AAT at 12 months (at the end of therapy)
Symptom Checklist-90-Revised (SCL-90R) | Change from baseline in SCL-90R at 12 months (at the end of therapy)
Stress Index for Parents of Adolescents (SIPA) | Change from baseline in SIPA at 12 months (at the end of therapy)
Stress Index for Parents of Adolescents (SIPA) | Change from baseline in SIPA at 18 months (follow-up)
drop-out rates | after 12 months (at the end of therapy)
cost-effectiveness | after 12 months (at the end of therapy)
  Cost-effectiveness will be measured by participation in training/school, rehospitalization, internment

OTHER OUTCOMES:
Working Alliance Inventory (WAI) | Change from baseline in WAI at 6 months
  Treatment related variable (moderator)
Working Alliance Inventory (WAI) | Change from baseline in WAI at 12 months (at the end of therapy)
  Treatment related variable (moderator)
Experiences in Close Relationships - Revised (ECR-R) | Change from baseline in ECR-R at 12 months (at the end of therapy)
  Treatment related variable (moderator)
Emotion Regulation Questionnaire (ERQ) | Change from baseline in ERQ at 12 months (at the end of therapy)
  Treatment related variable (moderator)
Emotion Regulation Questionnaire (ERQ) | Change from baseline in ERQ at 18 months (follow-up)
  Treatment related variable (moderator)
Zurich Brief Questionnaire for the Assessment of Parental Behaviors (ZKE) | Change from baseline in ZKE at 12 months (at the end of therapy)
  Treatment related variable (moderator)
The Mini-International Neuropsychiatric Interview (MINI) | Change from baseline in MINI at 12 months (at the end of therapy)
  Treatment related variable (moderator)
Youth Psychopathy Traits Inventory (YPI) | only baseline assessment
  Treatment related variable (moderator)
Cultural-Fair-Test (CFT-2) | only baseline assessment
  Treatment related variable (moderator)
Childhood Experience of Care and Abuse Questionnaire (CECA-Q) | only baseline assessment
  Treatment related variable (moderator)
Dimensional Assessment of Personality Pathology - Basic Questionnaire (DAPP-BQ) | only baseline assessment
  Treatment related variable (moderator)

CONTACTS AND LOCATIONS:
Overall Officials: Svenja Taubner, Prof., Principal Investigator — Institute for Psychosocial Prevention, Heidelberg University
Locations (1):
- Heidelberg University, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Taubner S, Zimmermann L, Ramberg A, Schroder P. Mentalization Mediates the Relationship between Early Maltreatment and Potential for Violence in Adolescence. Psychopathology. 2016;49(4):236-246. doi: 10.1159/000448053. Epub 2016 Aug 23. PMID 27548462
- [Background] Rossouw TI, Fonagy P. Mentalization-based treatment for self-harm in adolescents: a randomized controlled trial. J Am Acad Child Adolesc Psychiatry. 2012 Dec;51(12):1304-1313.e3. doi: 10.1016/j.jaac.2012.09.018. PMID 23200287
- [Background] Taubner S, White LO, Zimmermann J, Fonagy P, Nolte T. Attachment-related mentalization moderates the relationship between psychopathic traits and proactive aggression in adolescence. J Abnorm Child Psychol. 2013 Aug;41(6):929-38. doi: 10.1007/s10802-013-9736-x. PMID 23512713
- [Background] McGauley G, Yakeley J, Williams W, Bateman AW. Attachment, mentalization and antisocial personality disorder. The possible contribution of mentalization-based treatment. European Journal of Psychotherapy & Counselling. 2011; 13 (4): 371-393; doi: 10.1080/13642537.2011.629118.
- [Derived] Hauschild S, Kasper L, Volkert J, Sobanski E, Taubner S. Mentalization-based treatment for adolescents with conduct disorder (MBT-CD): a feasibility study. Eur Child Adolesc Psychiatry. 2023 Dec;32(12):2611-2622. doi: 10.1007/s00787-022-02113-4. Epub 2022 Nov 25. PMID 36434148
- [Derived] Taubner S, Hauschild S, Kasper L, Kaess M, Sobanski E, Gablonski TC, Schroder-Pfeifer P, Volkert J. Mentalization-based treatment for adolescents with conduct disorder (MBT-CD): protocol of a feasibility and pilot study. Pilot Feasibility Stud. 2021 Jul 2;7(1):139. doi: 10.1186/s40814-021-00876-2. PMID 34215323